CLINICAL TRIAL: NCT00956111
Title: A Double-blind, Randomized, Stratified and Controlled Clinical Trial With Split-virion and Whole-virion, Adjuvanted and Non-adjuvanted Influenza A/H1N1 Vaccines in Healthy Adults, Elders, Adolescents and Children
Brief Title: A Clinical Trial With Influenza A/H1N1 Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PanFlu-4001
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2009-10

CONDITIONS: Influenza
Keywords: Novel Influenza A/H1N1 Vaccine; Immunogenictiy; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- split-virion, adjuvanted H1N1 vaccine of 7.5 μg (Experimental): 300 participants (100 adults, 100 adolescents and 100 children) to receive split-virion, adjuvanted H1N1 vaccine of 7.5 μg on day 0 and 21.
  Interventions: Biological: split-virion, adjuvanted H1N1 vaccine of 7.5 μg per dose
- split-virion, adjuvanted H1N1 vaccine of 15 μg (Experimental): 300 participants (100 adults, 100 adolescents and 100 children) to receive split-virion, adjuvanted H1N1 vaccine of 15 μg on day 0 and 21.
  Interventions: Biological: split-virion, adjuvanted H1N1 vaccine of 15 μg per dose
- split-virion, non-adjuvanted H1N1 vaccine of 15 μg (Experimental): 300 participants (100 adults, 100 adolescents and 100 children) to receive split-virion, non-adjuvanted H1N1 vaccine of 15 μg on day 0 and 21.
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg per dose
- split-virion, non-adjuvanted H1N1 vaccine of 30 μg (Experimental): 300 participants (100 adults, 100 adolescents and 100 children) to receive split-virion, non-adjuvanted H1N1 vaccine of 30 μg on day 0 and 21.
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 30 μg per dose
- whole-virion, adjuvanted H1N1 vaccine of 5 μg (Experimental): 100 adults to receive whole-virion, adjuvanted H1N1 vaccine of 5 μg on day 0 and 21.
  Interventions: Biological: whole-virion, adjuvanted H1N1 vaccine of 5 μg per dose
- whole-virion, adjuvanted H1N1 vaccine of 10 μg (Experimental): 200 participants: 100 adults to receive whole-virion, adjuvanted H1N1 vaccine of 10 μg on day 0 and 21.
  100 elders to receive whole-virion, adjuvanted H1N1 vaccine of 10 μg on day 0 only.
  Interventions: Biological: whole-virion, adjuvanted H1N1 vaccine of 10 μg per dose
- Placebo control (Placebo Comparator): 100 adults to receive placebo control (Phosphate Buffer Saline) on day 0 and 21.
  Interventions: Biological: placebo control

INTERVENTIONS:
Biological: split-virion, adjuvanted H1N1 vaccine of 7.5 μg per dose — 100 adults, 100 adolescents and 100 children were assigned to receive 2 doses of 7.5μg split-virion, adjuvanted H1N1 vaccine 21 days apart.
  Arms: split-virion, adjuvanted H1N1 vaccine of 7.5 μg
Biological: split-virion, adjuvanted H1N1 vaccine of 15 μg per dose — 100 adults, 100 adolescents and 100 children were assigned to receive 2 doses of 15μg split-virion, adjuvanted H1N1 vaccine 21 days apart.
  Arms: split-virion, adjuvanted H1N1 vaccine of 15 μg
Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg per dose — 100 adults, 100 adolescents and 100 children were assigned to receive 2 doses of 15μg split-virion, non-adjuvanted H1N1 vaccine 21 days apart.
  Arms: split-virion, non-adjuvanted H1N1 vaccine of 15 μg
Biological: split-virion, non-adjuvanted H1N1 vaccine of 30 μg per dose — 100 adults, 100 adolescents and 100 children were assigned to receive 2 doses of 30μg split-virion, non-adjuvanted H1N1 vaccine 21 days apart.
  Arms: split-virion, non-adjuvanted H1N1 vaccine of 30 μg
Biological: whole-virion, adjuvanted H1N1 vaccine of 5 μg per dose — 100 adults were assigned to receive 2 doses of 5μg whole-virion, adjuvanted H1N1 vaccine 21 days apart.
  Arms: whole-virion, adjuvanted H1N1 vaccine of 5 μg
Biological: whole-virion, adjuvanted H1N1 vaccine of 10 μg per dose — 100 adults were assigned to receive 2 doses of 10μg whole-virion, adjuvanted H1N1 vaccine 21 days apart. 100 elders were assigned to receive 1 doses of 10μg whole-virion, adjuvanted H1N1 vaccine
  Arms: whole-virion, adjuvanted H1N1 vaccine of 10 μg
Biological: placebo control — 100 adults were assigned to receive 2 doses of placebo 21 days apart.
  Arms: Placebo control

SUMMARY:
A single center, stratified, randomized and double-blind phase IV clinical trial is to be conducted in healthy elders (equal to or more than 61 years), adults (18-60 years), adolescents (12-17 years) and children (3-11 years) to evaluate the safety and immunogenicity of Sinovac's split-virion or whole-virion novel influenza A (H1N1) vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female aged 3 and older
2. Be able to show legal identity card for the sake of recruitment
3. Volunteers or their guardians are able to understand and sign the informed consent

Exclusion Criteria:

1. Cases, cured cases and close contact of influenza A (H1N1) virus
2. Women of pregnancy, lactation or about to be pregnant in 60 days
3. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
4. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
5. Autoimmune disease or immunodeficiency
6. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
7. Diabetes mellitus (type I or II), with the exception of gestational diabetes
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
10. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
11. Active malignancy or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study
12. Seizure disorder other than:

    * Febrile seizures under the age of two years old
    * Seizures secondary to alcohol withdrawal more than 3 years ago, or
    * A singular seizure not requiring treatment within the last 3 years
13. Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen
14. Guillain-Barre Syndrome
15. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
16. History of any blood products or seasonal influenza vaccine administration within 3 months before the dosing
17. Administration of any other investigational research agents within 30 days before the dosing
18. Administration of any live attenuated vaccine within 30 days before the dosing
19. Administration of subunit or inactivated vaccines, e.g., pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
20. Be receiving anti-TB prophylaxis or therapy currently
21. Axillary temperature > 37.0 centigrade at the time of dosing
22. Psychiatric condition that precludes compliance with the protocol:

    * Past or present psychoses
    * Past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years
    * Disorder requiring lithium
    * Suicidal ideation occurring within five years prior to enrollment
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1614 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evaluate immunogenicity and safety of influenza A （H1N1）vaccines in elders, adults, adolescent and children . | July 2009- Sept. 2009

SECONDARY OUTCOMES:
Provide a basis to determine the best type and dose of vaccine and immunization procedures | July 2009- Sept. 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Centers for Diseases Control and Prevention, Beijing, China

REFERENCES:
- [Derived] Wu J, Li W, Wang HQ, Chen JT, Lv M, Zhou JC, Liang XF, Fang HH, Liu Y, Liu LY, Wang X, Zhang WL, Zhang XM, Song LF, Qiu YZ, Li CG, Wang JZ, Wang Y, Yin WD. A rapid immune response to 2009 influenza A(H1N1) vaccines in adults: a randomized, double-blind, controlled trial. J Infect Dis. 2010 Sep 1;202(5):675-80. doi: 10.1086/655226. PMID 20632888
- [Derived] Liang XF, Wang HQ, Wang JZ, Fang HH, Wu J, Zhu FC, Li RC, Xia SL, Zhao YL, Li FJ, Yan SH, Yin WD, An K, Feng DJ, Cui XL, Qi FC, Ju CJ, Zhang YH, Guo ZJ, Chen PY, Chen Z, Yan KM, Wang Y. Safety and immunogenicity of 2009 pandemic influenza A H1N1 vaccines in China: a multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2010 Jan 2;375(9708):56-66. doi: 10.1016/S0140-6736(09)62003-1. Epub 2009 Dec 15. PMID 20018364